CLINICAL TRIAL: NCT04700228
Title: Comparison of Doses of Dexmedetomidine With Bupivacaine in Caudal Block for Duration of Analgesia in Paediatric Infraumblical Surgeries.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dr. Ruth K.M. Pfau Civil Hospital, Karachi (Other Government)
Responsible Party: Principal Investigator, Haris Chohan, Faculty Member, Dr. Ruth K.M. Pfau Civil Hospital, Karachi
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Haris123
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Pain, Postoperative
Keywords: Postoperative pain; Regional Anaesthesia; Caudal Block; Dexmedetomidine; Infraumbilical surgeries
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Factorial Assignment Anesthesia will be induced with 100% oxygen and sevoflurane 8%. Once achieving the desired depth of anesthesia, I/V access will be taken. Propofol 3mg/kg and Nalbuphine 0.1mg/kg will be given. LMA of desirable size will be placed. After this, patient would be placed in lateral position for caudal Block. After all aseptic measures, Caudal Block procedure will be done with help of 23G needle by anatomical landmarks. On negative aspiration of the syringe, one of the drug combinations as explained under 'arms and intervention' will be used for the caudal block. First surgical incision will be given 10 mins after the application of caudal block. After the completion of surgery, LMA will be removed once the patient is awake and the patient will be shifted to PACU. IV paracetamol 15mg/kg will be given if FLACC score is more than 4 at any point during the surgery.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (Placebo Comparator): 0.25% bupivacaine at a total volume of 0.5ml/kg.
  Interventions: Drug: Bupivacaine Hydrochloride
- Group BD1 (Active Comparator): 0.25% bupivacaine + 1mcg/kg dexmedetomidine at a total volume of 0.5ml/kg.
  Interventions: Drug: Bupivacaine Hydrochloride; Drug: Dexmedetomidine
- Group BD2 (Active Comparator): 0.25% bupivacaine + 0.5mcg/kg dexmedetomidine at a total volume of 0.5ml/kg.
  Interventions: Drug: Bupivacaine Hydrochloride; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — We are going to see the effects of dexmedetomidine as an adjunct to bupivacaine in caudal block. In first (control) group (group C) only bupivacaine will be given. Group BD1 patients will be given bupivacaine plus 1mcg/kg dexmedetomidine. Group BD2 patients will get bupivacaine plus 0.5mcg/kg dexmedetomidine. All the groups will be given a volume of 0.5ml/kg.
Drug: Dexmedetomidine — We are going to see the effects of dexmedetomidine as an adjunct to bupivacaine in caudal block. In first (control) group (group C) only bupivacaine will be given. Group BD1 patients will be given bupivacaine plus 1mcg/kg dexmedetomidine. Group BD2 patients will get bupivacaine plus 0.5mcg/kg dexmedetomidine. All the groups will be given a volume of 0.5ml/kg.
  Arms: Group BD1; Group BD2

SUMMARY:
Various methods are used to control post-operative pain among children. Amongst these methods, caudal block is one of the most favoured, prominent and dependable methods for providing reliable analgesia in surgeries below umbilicus.

This study is to compare two doses of Dexmedetomidine added as adjunct to local anaesthesia using reduced dose in caudal block for prolonging the duration of analgesia. Our secondary outcomes will include blood pressure, heart rate, urinary retention, nausea and vomiting in the paediatric population.

DETAILED DESCRIPTION:
Pain is one the most underrated, misunderstood and often underdiagnosed field especially in children. Pain is an unpleasant feeling which is basically a subjective feeling, which in children is poorly expressed. Failure to control pain during childhood ultimately results in having chronic adverse effects which include altered sleep, eating habits and neuroendocrine responses and increased sensitivity to pain in the following pain episodes.

Successful postoperative pain management is one of the main pillars of anaesthesia. Regional Anaesthesia has gained a lot of popularity over the past few years in paediatrics. Approximately one-quarter of analgesic procedures currently performed on children are done by regional analgesic techniques. There are various methods that are being currently used to control post-operative pain among children. Amongst these methods, caudal block is one of the most favoured, prominent and dependable methods for providing reliable analgesia in surgeries below umbilicus. However, it has a drawback of being having a limited time of action when used as a single shot technique. This time limit can be increased significantly by the addition of different adjuvants along with local anaesthetic drugs in caudal block, which not only helps the anaesthesiologist in giving a better quality of anaesthesia and analgesia but it leads up to creating a desirable intraoperative environment for the surgeon as well. Better control over intraoperative and post-operative analgesia also helps the anaesthesiologist in giving reduced levels of anaesthesia which caused reduced amount of postoperative sedation as well.

Dexmedetomidine has a specific affinity for α2-adrenoreceptor having sedative and analgesic properties, which makes it an ideal adjuvant agent. The landmark ability of this adjuvant is that it causes minimal respiratory depression even at high dosages. A number of studies have been done until now that have proved successfully that dexmedetomidine can be used as an adjuvant in caudal block, in children, in enhancing post-operative analgesia. Although there is insufficient data available, various studies have demonstrated the dose of dexmedetomidine in Caudal Block ranging from 0.5 µg/kg to 2 µg/kg. According to an up to date review anaesthesia will last longer with dexmedetomidine as compared to morphine when used, as haemodynamics were found to be stable mostly when dexmedetomidine was used. However bradycardia was mostly related to a dose of 2 mcg/kg of dexmedetomidine. A study published in 2019 documented a decrease in heart rate, not requiring active management, in the dexmedetomidine group at a dose of 1mcg/kg.

Our objective is to compare two doses of Dexmedetomidine added as adjunct to local anaesthesia using reduced dose in caudal block for prolonging the duration of analgesia. Our secondary outcomes will include blood pressure, heart rate, urinary retention, nausea and vomiting in the paediatric population.

Patient meeting inclusion criteria visiting paediatric operating room will be inducted in the study. Informed and written consent will be taken from parents/guardian explained about the potential risk and benefits of study. Patients' demographic details like age, sex, and weight will be collected by filling the relevant proforma. A total of 162 patients will be divided into three equal groups randomly by lottery method. The observer and the anaesthesiologist who will induce the patient will be blinded regarding the group in which the patient will be placed.

Pre operatively, a detailed history, examination and related laboratory investigations will be seen as a part of hospital pre-operative assessment protocol. On arrival to operation theatre, monitors (SpO2, Pulse Oximeter, NIBP, pre cordial stethoscope and ECG) will be applied. Emergency drugs will be prepared already before the patient arrives in operation theatre. Anaesthesia will be induced with 100% oxygen and sevoflurane 8% using Jackson Rees Circuit. Once the desired depth of anaesthesia is achieved, I/V access will be taken. Propofol 3mg/kg and Nalbuphine 0.1mg/kg will be given and Sevoflurane will be set at 3%. LMA of desirable size will be placed. After this, patient would be placed in lateral position. Sufficient exposure would be done for Caudal Block. After taking all aseptic measures, Caudal Block procedure will be done with help of 23G needle after identifying the anatomical landmarks. Correction position of the needle will be confirmed by swoosh and whoosh test. On aspiration of the syringe if it is negative for CSF and blood, then one of the following drug combinations will be used for the caudal block.

Group C (control): 0.25% bupivacaine at a total volume of 0.5ml/kg Group BD1: 0.25% bupivacaine + 1mcg/kg dexmedetomidine at a total volume of 0.5ml/kg Group BD2: 0.25% bupivacaine + 0.5mcg/kg dexmedetomidine at a total volume of 0.5ml/kg After dressing the injection site, the patient will be turned supine. Vitals of the patient including heart rate, blood pressure, SpO2 and respiratory will be recorded before the induction of caudal block and there after every 10 minutes. Inadequate analgesia or unsuccessful block will be labelled if there would be a 20% increase in heart rate of the patient as compared to the baseline recording. If the caudal block is insufficient that case will not be included in the study. Hypotension and bradycardia will be recorded and treated with fluid bolus and atropine respectively. . The first surgical incision would be given 10 mins after the application of caudal block. After the completion of the surgery, inhalation gas will be closed and patient will be given 100% oxygen only. LMA will be removed once the patient is awake and the patient will be shifted to Post Anaesthesia Care Unit (PACU). Here patient's vitals will be monitored and pain will be assessed at 1, 2, 4, 6 and 12 hours after the application of caudal block using FLACC scale16. Time taken for the requirement of first rescue analgesia will also be recorded. Intravenous paracetamol 15mg/kg will be given if FLACC score is more than 4 at any of the above mentioned time. Secondary findings like heart rate, blood pressure, respiratory depression, urinary retention, nausea and vomiting will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) Status I and II
* Aged between 1 to 6 years
* Planned for below umbilicus elective surgery

Exclusion Criteria:

* Refusal to consent by parent/guardian
* Injection site infection
* Coagulation disorders
* Congenital abnormalities of lower spine and meninges
* Anticipated difficult airway requiring endotracheal intubation and intermittent positive pressure ventilation
* Prone position surgical procedures
* Known drug allergy history

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Duration of Analgesia | 1 hour after caudal block
  Time period between administration of block until the time face, legs, activity, cry, consolability (FLACC) score reached ≥4
Duration of Analgesia | 2 hours after caudal block
  Time period between administration of block until the time face, legs, activity, cry, consolability (FLACC) score reached ≥4
Duration of Analgesia | 4 hours after caudal block
  Time period between administration of block until the time face, legs, activity, cry, consolability (FLACC) score reached ≥4
Duration of Analgesia | 6 hours after caudal block
  Time period between administration of block until the time face, legs, activity, cry, consolability (FLACC) score reached ≥4
Duration of Analgesia | 12 hours after caudal block
  Time period between administration of block until the time face, legs, activity, cry, consolability (FLACC) score reached ≥4

SECONDARY OUTCOMES:
Heart Rate (bradycardia) | 1 hour after caudal block.
  heart rate less than 60 beats/min for ages above 1 year.
Heart Rate (bradycardia) | 2 hours after caudal block.
  heart rate less than 60 beats/min for ages above 1 year.
Heart Rate (bradycardia) | 4 hours after caudal block.
  heart rate less than 60 beats/min for ages above 1 year.
Heart Rate (bradycardia) | 6 hours after caudal block.
  heart rate less than 60 beats/min for ages above 1 year.
Heart Rate (bradycardia) | 12 hours after caudal block.
  heart rate less than 60 beats/min for ages above 1 year.
Blood Pressure | 1 hour after caudal block.
  Decrease in systolic blood pressure < 25% from the baseline
Blood Pressure | 2 hours after caudal block.
  Decrease in systolic blood pressure < 25% from the baseline
Blood Pressure | 4 hours after caudal block.
  Decrease in systolic blood pressure < 25% from the baseline
Blood Pressure | 6 hours after caudal block.
  Decrease in systolic blood pressure < 25% from the baseline
Blood Pressure | 12 hours after caudal block.
  Decrease in systolic blood pressure < 25% from the baseline
Postoperative Respiratory Depression | 1 hour after caudal block.
  if the SpO2 is less than 95% or breathing rate is less than 10 breaths per minute.
Postoperative Respiratory Depression | 2 hours after caudal block.
  if the SpO2 is less than 95% or breathing rate is less than 10 breaths per minute.
Postoperative Respiratory Depression | 4 hours after caudal block.
  if the SpO2 is less than 95% or breathing rate is less than 10 breaths per minute.
Postoperative Respiratory Depression | 6 hours after caudal block.
  if the SpO2 is less than 95% or breathing rate is less than 10 breaths per minute.
Postoperative Respiratory Depression | 12 hours after caudal block.
  if the SpO2 is less than 95% or breathing rate is less than 10 breaths per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Haris Chohan, FCPS Pakistan, Principal Investigator — Dr. Ruth KM Pfau Civil Hospital, Dow University of Health Sciences Karachi, Pakistan; Syed Farjad Sultan, FCARCSI, PhD, Principal Investigator — Dr. Ruth KM Pfau Civil Hospital, Dow University of Health Sciences Karachi, Pakistan; Arun Kumar, FCPS, Principal Investigator — Dr. Ruth KM Pfau Civil Hospital, Dow University of Health Sciences, Karachi, Pakistan
Locations (1):
- Dr. Haris Chohan, Karachi, Sindh, Pakistan